CLINICAL TRIAL: NCT00651378
Title: An Open-Label, Randomized, Parallel-Group, Multicenter Study to Compare the Efficacy and Safety of "Switching" to Rosuvastatin 10 mg Daily Versus Atorvastatin 10 mg Daily With Ezetimibe 10 mg Daily Versus Doubling the Dose of Atorvastatin to 20 mg Daily in Subjects With Hypercholesterolemia and Atherosclerotic or Coronary Vascular Disease or Diabetes Mellitus Who Have Not Achieved Study Target LDL-C Goal While Dosing With Atorvastatin 10 mg Daily
Brief Title: Switching to Rosuvastatin Versus Adding Ezetimibe to Atorvastatin Versus Doubling the Dose of Atorvastatin in Patients With Hypercholesterolemia and Risk Factors (P03708)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment [HIGH SCREEN FAILURE RATE]
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03708
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Coronary Artery Disease | interventions — Rosuvastatin Calcium; Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin
- Ezetimibe + Atorvastatin (Active Comparator)
  Interventions: Drug: Ezetimibe + Atorvastatin
- Double Atorvastatin (Active Comparator)
  Interventions: Drug: Double Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — oral tablets: rosuvastatin 10 mg once daily for 6 weeks (switch from previous run-in with atorvastatin 10 mg daily)
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Ezetimibe + Atorvastatin — oral tablets: ezetimibe 10 mg plus atorvastatin 10 mg once daily for 6 weeks (add ezetimibe to previous run-in with atorvastatin 10 mg daily)
  Other Names: SCH 58235; Zetia; Lipitor
  Arms: Ezetimibe + Atorvastatin
Drug: Double Atorvastatin — oral tablets: atorvastatin 20 mg once daily for 6 weeks (double dose from previous run-in with atorvastatin 10 mg daily)
  Other Names: Lipitor
  Arms: Double Atorvastatin

SUMMARY:
This study assesses whether adding ezetimibe 10 mg/d to ongoing treatment with atorvastatin 10 mg/d is more effective than switching the subject to treatment with rosuvastatin 10 mg/d or doubling the dose of atorvastatin to 20 mg/d is more effective in achieving goal LDL-cholesterol of <2.5 mmol/L. Treatment phase is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years of age;
* Stabilized on atorvastatin 10 mg daily and by subject reported history had taken at least 80% of daily doses for the 4 weeks preceding Visit 1;
* LDL-C concentration greater than or equal to 2.5 mmol/L to less than or equal to 160 mg/dL (less than or equal to 4.1 mmol/L) based on blood specimens taken at Visit 1, using the Friedewald calculation as described in the Protocol,Section 8.8. (The lipid profiles at Visit 3 (baseline) and all subsequent visits were kept "blinded" until data analysis);
* Triglyceride concentration of less than 350 mg/dL (less than 3.99 mmol/L) based on blood specimens taken at Visit 1;
* Documented atherosclerotic disease, CHD, or diabetes mellitus;
* Liver transaminases (ALT, AST) less than 50% above the upper limit of normal, with no active liver disease, and CPK less than 50% above the upper limit of normal as tested in blood specimens taken at Visit 1;
* Clinical laboratory tests (CBC, blood chemistries, urinalysis) taken at Visit 1 must have been within normal limits or clinically acceptable to the Investigator;
* Had been previously prescribed a cholesterol lowering diet and exercise program at least 4 weeks prior to Visit 1 and had been advised to continue the same diet and exercise program during the study;
* Reported a stable weight history for at least 4 weeks prior to randomization at Visit 3 (baseline visit);
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and willing to continue the same regimen for the duration of the study;
* Women of childbearing potential (included women who were less than 1 year postmenopausal and women who became sexually active) must have been using an acceptable method of birth control (for example, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or been surgically sterilized (for example, hysterectomy or tubal ligation).
* Free of any clinically significant diseases other than hyperlipidemia, CHD, or diabetes mellitus that would interfere with study evaluations;
* Understood and were able to adhere to the dosing and visit schedules, and demonstrated their willingness to participate in the study and comply with its procedures by signing a written informed consent.

Exclusion Criteria:

* Consumption greater than 14 alcoholic drinks per week. (A drink is: a can of beer [1/2 pint or 250 ml], glass of wine, or single measure of spirits);
* Any condition or situation which, in the opinion of the Investigator, might have posed a risk to the subject or interfered with participation in the study;
* Body mass index (BMI) >= 35 Kg/m^2 at Visit 2 (Screening);
* Women who were pregnant or nursing;
* Failure to observe the designated washout periods for any of the prohibited medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2004-09-01 (Actual); Primary Completion 2005-06-01 (Actual); Study Completion 2005-06-01 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C level from baseline to the study endpoint. | 6 weeks

SECONDARY OUTCOMES:
Percent changes from baseline to the end of treatment in the concentrations of total cholesterol (TC), non-HDL-C, apo B, triglycerides (TG), HDL-C, LDL-C/HDL-C ratio, and TC/HDL-C ratio. | 6 weeks
Adverse events, laboratory test results, vital signs. | Throughout study